CLINICAL TRIAL: NCT01998542
Title: Phase II Study Designed To Evaluate Safety and Tumor Debulking Mechanism of an Individualized Cancer Vaccine (AllovaxTM) in Patients With Metastatic or Recurrent Cancer of the Head and Neck.
Brief Title: Safety and Tolerability Study of AlloVax(TM) in Patients With Metastatic or Recurrent Cancer of the Head and Neck
Acronym: HNC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-010-HNC
Record Dates: First submitted 2013-11-21; First posted 2013-11-29 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2016-08

CONDITIONS: Cancer of Head and Neck; Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and neck cancers; tumor vaccine; immunotherapy; personalized anti-cancer vaccine
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: 12 subjects with externally measurable disease
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AlloStim+CRCL (Experimental): AlloStim priming followed by AlloStim+CRCL priming and AlloStim IV. 3 cycles
  Interventions: Biological: AlloVax; Biological: CRCL; Biological: AlloStim

INTERVENTIONS:
Biological: AlloVax — Personalized anti-cancer vaccine with AlloStim(TM) and CRCL
  Other Names: CRCL and AlloStim
Biological: CRCL — autologous tumor-derived chaperone protein mixture
  Other Names: Chaperone Rich Cell Lysate; CRCL injection
Biological: AlloStim — AlloStim (ID) injection AlloStim (IV) infusion
  Other Names: AlloStim ID; AlloStim IV

SUMMARY:
The purpose of this study is to determine the safety and tumor debulking efficacy of personalized anti-cancer vaccine AlloVax(TM) in Subjects with confirmed recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) who cannot be treated with surgery, chemotherapy or radiation. AlloVax(TM) is a personalized anti-cancer vaccine combining Chaperone Rich Cell Lysate (CRCL) as a source of tumor antigen prepared from patient's tumor and AlloStim(TM) as an adjuvant. The combination of CRCL and AlloStim(TM) is designed to provide cross-reactivity of alloantigen specific recognition with tumor-specific recognition. All the key components necessary to develop tumor-specific immunity by creating the inflammatory environment necessary to overcome the HNC immunosuppressive environment, breaking tumor immune tolerance, and provision of specific HNC antigens for generation of a specific adaptive anti-tumor response.

DETAILED DESCRIPTION:
This is a Phase II study following up on a previous Phase I/II study in chemotherapy refractory metastatic disease with <90 day survival expectancy. In the Phase I/II study all patients progressed using RECIST criteria. However, 11/42 (26%) were alive at 1yr and 9/42 (21%) alive at 2 yr. Therefore, CT scans did not correlate with clinical presentation and "pseudo-progression" was suspected. This study was designed to select subjects with visible tumor burden on the head, neck or tongue that could be measured and photographed so as not to rely solely on CT scans to determine anti-tumor debulking efficacy. Subjects are initially primed with intradermal AlloStim(TM) injections creating systemic anti-allo-specific cellular immunity. Tumor biopsy samples taken prior to dosing were processed into personalized Chaperone Rich Cell Lysate (CRCL) vaccine containing enriched heat shock proteins which are believed to chaperone tumor-specific neoantigens . AlloStim(TM) was then injected with CRCL into primed subjects to create tumor-specific cellular immunity. Subsequently, subjects are infused with intravenous AlloStim(TM) to cause extravasation of memory cells to the tumor lesions. The protocol including intradermal AlloStim(TM) day 0, 3, 7, 10. Intradermal AlloStim(TM)+CRCL on days 14, 17, 21, 24. Intravenous AlloStim(TM) day 28. This experimental treatment schedule will continue for 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and female patients aged 18 to 70 years old, inclusive, at screening visit.
2. Patients with histopatholologically or cytologically confirmed diagnosis of recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) that is incurable with surgery, chemotherapy or radiation. No nasopharyngeal primaries.
3. Patients must have a tumor safely accessable for biopsy resulting in a minimum of 0.1 g of tumor sample for CRCL processing.
4. Patients must have visible external tumors measurable with at least one lesion deemed to be safely accessible for serial biopsy.
5. ECOG ≤2.
6. The result of screening test were in the criteria:

   6.1 Adequate organ function including:

   A. Marrow:
   * WBC >3000/mm3
   * Platelets >100,000/mm3.
   * Absolute neutrophil count ≥ 1,500/mm³
   * Hemoglobin ≥ 10.0 g/dL (transfusion allowed)

   B. Hepatic:
   * Serum Total bilirubin < 2 x ULN mg/dL,
   * ALT (SGPT) / AST (SGOT) ≤3 x upper limit of normal (ULN).

   C. Renal:
   * Serum creatinine (SCR) <2.0 x ULN, or
   * Creatinine clearance (CCR) >30 mL/min.

   6.2 All patients have a pre-study echocardiogram without significant abnormalities or Ejection fraction >50%.

   6.3 All patients must be screened to be negative for HIV1, HIV2, HTLVI, HTLVII, HBV, HCV and RPR (syphilis).

   6.4 Women of child-bearing potential must have a negative urine or serum pregnancy test result within 72 hours prior to the start of study drug administration.
7. All patients of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product.
8. Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate.

Exclusion Criteria:

1. Clinical evidence or radiological evidence of nasopharyngeal primaries.
2. Clinical evidence or radiological evidence of brain metastasis.
3. History of severe hypersensitivity to monoclonal antibody drugs or any contraindication to any of the study drugs.
4. Concomitant active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis).
5. Prior experimental therapy or cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine).
6. Clinical requirement for systemic steroids or current immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 1 month of study entry.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, requiring parenteral antibiotics, symptomatic congestive heart failure, severe myocardial insufficiency, cardiac arrhythmia
8. All infections must be resolved and the patient must remain a febrile for seven days prior to being placed in the study.
9. History of blood transfusion reactions.
10. Psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation.
11. Pregnant or breast feeding.

The patient will discontinuation from the participation in the study:

1. Less than 12 doses of CRCL able to be produced
2. Tumor sample for CRCL processing contains less than 80% tumor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Tumor Response | baseline, every 28 days for 5 months (CT scan confirmation at baseline and day 90 and day 150)
  Tumor response evaluation by clinical exam including photographs of visible tumor lesions on head, neck and/or tongue (endoscopic) and by CT scan assessment for change in target lesion tumor volume (TV). TV is defined as the volume occupied by macroscopic visible target lesion in two longest cross-sectional diameters.

SECONDARY OUTCOMES:
Anti-tumor immune response | baseline, 30 days after the last dose
  change in tumor pathology and immune cell inflitration
Anti-Tumor Response | baseline and 30 days after the last dose
  expression of CTLA4.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Har-Noy, Dr., Study Director — Mirror Biologics, Inc.
Locations (1):
- National Cancer Institute of Thailand, Bangkok, Thailand

REFERENCES:
- [Result] Epple LM, Bemis LT, Cavanaugh RP, Skope A, Mayer-Sonnenfeld T, Frank C, Olver CS, Lencioni AM, Dusto NL, Tal A, Har-Noy M, Lillehei KO, Katsanis E, Graner MW. Prolonged remission of advanced bronchoalveolar adenocarcinoma in a dog treated with autologous, tumour-derived chaperone-rich cell lysate (CRCL) vaccine. Int J Hyperthermia. 2013 Aug;29(5):390-8. doi: 10.3109/02656736.2013.800997. Epub 2013 Jun 20. PMID 23786302
- [Result] Mayer-Sonnenfeld T, Har-Noy M, Lillehei KO, Graner MW. Proteomic analyses of different human tumour-derived chaperone-rich cell lysate (CRCL) anti-cancer vaccines reveal antigen content and strong similarities amongst the vaccines along with a basis for CRCL's unique structure: CRCL vaccine proteome leads to unique structure. Int J Hyperthermia. 2013 Sep;29(6):520-7. doi: 10.3109/02656736.2013.796529. Epub 2013 Jun 4. PMID 23734882
- [Result] LaCasse CJ, Janikashvili N, Larmonier CB, Alizadeh D, Hanke N, Kartchner J, Situ E, Centuori S, Har-Noy M, Bonnotte B, Katsanis E, Larmonier N. Th-1 lymphocytes induce dendritic cell tumor killing activity by an IFN-gamma-dependent mechanism. J Immunol. 2011 Dec 15;187(12):6310-7. doi: 10.4049/jimmunol.1101812. Epub 2011 Nov 9. PMID 22075702
- [Result] Janikashvili N, LaCasse CJ, Larmonier C, Trad M, Herrell A, Bustamante S, Bonnotte B, Har-Noy M, Larmonier N, Katsanis E. Allogeneic effector/memory Th-1 cells impair FoxP3+ regulatory T lymphocytes and synergize with chaperone-rich cell lysate vaccine to treat leukemia. Blood. 2011 Feb 3;117(5):1555-64. doi: 10.1182/blood-2010-06-288621. Epub 2010 Dec 1. PMID 21123824
- [Result] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Result] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441
- See also: Cancer — http://www.nlm.nih.gov/medlineplus/cancer.html
- See also: Head and Neck Cancer — http://www.nlm.nih.gov/medlineplus/headandneckcancer.html